CLINICAL TRIAL: NCT04330859
Title: NEO Rehab Program for Premature Infants at Risk for Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Santina Zanelli, Associate Professor, Neonatology, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UVirginia; R03HD097727 (NIH)
Record Dates: First submitted 2019-04-29; First posted 2020-04-02 (Actual); Results first posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Cerebral Palsy; Prematurity; Early Intervention; Family Centered Care
Keywords: cerebral palsy; prematurity; early intervention; parent-driven; brain plasticity; motor outcome
MeSH Terms: conditions — Cerebral Palsy; Premature Birth

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Parent-driven intervention bundle of 6 evidence-based elements: vocal soothing, scent exchange, comforting touch, kangaroo care, infant massage and physical therapy
  Interventions: Other: NeoRehab Bundle
- Routine care (Placebo Comparator): Routine care per unit guidelines
  Interventions: Other: Routine care

INTERVENTIONS:
Other: NeoRehab Bundle — The NICU rehabilitation program includes six multimodal, GA appropriate, parent-administered interventions (vocal soothing, scent exchange, comforting touch, kangaroo care, infant massage and physical therapy)
  Arms: Intervention
Other: Routine care — Routine NICU care including talking, touching and holding the participant per unit guideline as well as physical therapy, occupational therapy, and speech therapy per unit guideline
  Arms: Routine care

SUMMARY:
The goal of this project is to investigate the acceptability, feasibility and fidelity of an innovative NICU rehabilitation program that will include six multimodal, gestational age (GA) appropriate, parent-administered interventions (vocal soothing, scent exchange, comforting touch, kangaroo care, infant massage and physical therapy). Using the general movement assessment (GMA) instrument, the investigators will determine the effects of this program on short-term motor outcomes (general movements (GMs), cranial nerves, posture, movements, tone, and reflexes) in premature infants (≤32 week's gestation and/or ≤1500 grams birthweight) identified as at-risk for CP. The short-term motor outcomes will be measured using the GMA, the Test of Infant Motor Performance (TIMP) and the Hammersmith Infant Neurological Examination (HINE) instruments. This novel program will be applied during the neonatal intensive care unit (NICU) hospitalization when the brain is highly plastic and actively developing with the goal to mitigate severity of brain injury and its impact on development.

DETAILED DESCRIPTION:
The two following specific aims will be tested:

Aim 1: Enroll 60 preterm infants (<32 weeks' gestation and/or ≤1500 grams) with abnormal GMA into a pilot randomized control trial to evaluate the acceptability, feasibility (practicality) and fidelity (adherence, exposure and engagement) of a multimodal GA appropriate rehabilitation program during NICU hospitalization compared to standard of care. The investigators will evaluate:

* Acceptability using recruitment, refusal, retention, and follow-up rates as well as weekly interviews with parental participants
* Feasibility (practicality) using direct observations and weekly interviews with parental participants
* Fidelity (adherence, exposure and engagement) using visitation data, activity logs, direct observations, and weekly interviews.

Aim 2: Examine the effect of a multimodal NICU-based rehabilitation program on short-term motor outcomes (general movements, cranial nerves, posture, movements, tone, and reflexes) of premature infants at risk for cerebral palsy (CP) at discharge from the NICU and at 3 months corrected age. The investigators hypothesize that this type of GA appropriate multimodal NICU-based rehabilitation program will positively impact short-term motor outcomes by normalizing general movements and improving TIMP and HINE scores.

ELIGIBILITY:
Inclusion Criteria:

* GA at birth: ≤32 weeks gestation and/or birthweight ≤1500 grams
* Infants 7 days or older
* Ability of parents or identified designated surrogate (e.g. grandparent) to perform the interventions
* Abnormal writhing GMs defined by the presence of a poor repertoire pattern on 2 consecutive assessments or the presence of a cramped-synchronized pattern on any assessment

Exclusion Criteria:

* Clinically unstable (requiring high frequency mechanical ventilation, vasopressor support, need for continuous intravenous pain or sedation medication)
* If their parents do not speak English
* If parental participation is hindered (e.g. incarceration).

Ages: 23 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2019-05-25 (Actual); Primary Completion 2020-10-10 (Actual); Study Completion 2021-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: santina zanelli, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Letzkus L, Conaway M, Miller-Davis C, Darring J, Keim-Malpass J, Zanelli S. A feasibility randomized controlled trial of a NICU rehabilitation program for very low birth weight infants. Sci Rep. 2022 Feb 2;12(1):1729. doi: 10.1038/s41598-022-05849-w. PMID 35110644

RESULTS

PARTICIPANT FLOW:
Groups:
- Parent-driven Multimodal Interventions: Parent-driven intervention bundle of 6 evidence-based elements: vocal soothing, scent exchange, comforting touch, kangaroo care, infant massage and physical therapy
  NeoRehab Bundle: The NICU rehabilitation program includes six multimodal, GA appropriate, parent-administered interventions (vocal soothing, scent exchange, comforting touch, kangaroo care, infant massage and physical therapy)
- Routine Care (Control Group): Routine care per unit guidelines
  Routine care: Routine NICU care including talking, touching and holding the participant per unit guideline as well as physical therapy, occupational therapy, and speech therapy per unit guideline
Period: Overall Study
Arm/Group | Parent-driven Multimodal Interventions | Routine Care (Control Group)
Started | 36 | 34
Completed | 25 | 26
Not Completed | 11 | 8

BASELINE CHARACTERISTICS:
Population: 70 patients consented and enrolled. Not all patients completed all portions of the studies resulting in different numbers for specific outcomes
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Routine Care | Total
Number analyzed (Participants) | 34 | 33 | 67
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 34 | 33 | 67
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: weeks] | 28.02 (2.70) | 28.75 (2.68) | 28.39 (2.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 10 | 24
  Male | 20 | 23 | 43
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black | 8 | 4 | 12
  Race: Caucasian | 26 | 29 | 55

OUTCOME MEASURES:

1. Primary Outcome: Acceptability
Description: The following measure will be used to measure study acceptability:
  % Recruitment rates during enrollment period
Time Frame: from day 1 of study screening through end of screening (approximately 1 year and3 months).
Measure: Count of Participants; unit: Participants
Groups:
- Study Acceptability: Acceptability of enrollment into study
Arm/Group | Study Acceptability
Number analyzed (Participants) | 99
Participants | 70

2. Primary Outcome: Retention Rates
Description: The following measure will be used to assess the retention rate of study participants:
  - Rate of follow-up at the 3 month outpatient visit
Time Frame: From discharge to 3 months follow-up
Measure: Number; unit: percentage of participants
Groups:
- Study Retention: Percent participant that remained in the study after enrollment
Arm/Group | Study Retention
Number analyzed (Participants) | 70
percentage of participants | 73

3. Primary Outcome: Adherence Rates
Description: Adherence rates were monitored by daily activity logs of interventions from enrollment day 1 to discharge for each visit day
Time Frame: from study enrollment (day 1) to study discharge
Measure: Number; unit: percentage of participants
Groups:
- Control: Routine care
Arm/Group | Intervention | Control
Number analyzed (Participants) | 32 | 33
percentage of participants | 0 | 0

4. Primary Outcome: Impact of the NeoRehab Bundle on Motor Performance Using the Test of Infant Motor Performance (TIMP)
Description: Motor outcomes will be assessed at NICU discharge and at 3 months using the Test of Infant Motor Performance (TIMP); 3 months outcome reported. TIMP score range = 0-142; lower scores indicate worse motor performance
Time Frame: 3 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention | Routine Care
Number analyzed (Participants) | 22 | 21
score on a scale | 86 [73 to 100] | 91 [83 to 99]

5. Primary Outcome: Impact of the NeoRehab Bundle on Neurologic Function as Assessed by the Hammersmith Infant Neurological Examination (HINE).
Description: Neurologic function will be assessed at NICU discharge and at 3 months postmenstrual age using the Hammersmith Infant Neurological Examination (HINE) instrument, 3 months outcome reported. The HINE is a 26 items scale that evaluates cranial nerve function, posture, quality and quantity of movements, muscle tone, and reflexes and reactions. Lower the score the poorer the motor function. HINE score range = 0-78 (with lower score indicating lower motor performance). The HINE has a sensitivity of 90% for prediction of motor outcome.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Routine Care
Number analyzed (Participants) | 25 | 26
score on a scale | 58.8 (7.2) | 57.2 (11.2)
Statistical Analysis 1: Comparison: Intervention; Test type: Superiority; p = 0.0543, t-test, 1 sided — 58.8 ± 7.2 (intervention) and 57.2 ± 11.2 (control; p = 0.0543); Agresti-Caffo = 95

6. Primary Outcome: Percent Abnormal General Movements
Description: The impact of the intervention on the infants' general movement will be assessed at NICU discharge and at 3 months postmenstrual age using the general movement assessment (GMA) tool. The GMA has been shown to reliably identify infants at high risk for CP and can be implemented shortly after birth making it an ideal screening tool for preterm infants. Cramped-synchronized writhing general movements followed by absent fidgety general movements is a movement pattern that has been shown to be highly specific of later development of cerebral palsy.
Time Frame: 3 months
Population: Abnormal general movements = absent fidgety classification
Measure: Number; unit: percentage of participants
Arm/Group | Intervention | Routine Care
Number analyzed (Participants) | 23 | 28
percentage of participants | 57 | 54

ADVERSE EVENTS:
Time Frame: from study enrollment (day 1) through study completion (approximately 2 years and 2 months)
Arm/Group | Intervention | Routine Care
All-Cause Mortality (participants affected / at risk) | 0/36 | 1/34
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/34
Other Adverse Events (participants affected / at risk) | 0/36 | 0/34

LIMITATIONS AND CAVEATS:
Lower than expected follow-up rates due to covid-19 restrictions

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-09-10): https://cdn.clinicaltrials.gov/large-docs/59/NCT04330859/Prot_SAP_000.pdf
  • Informed Consent Form (2019-04-23): https://cdn.clinicaltrials.gov/large-docs/59/NCT04330859/ICF_001.pdf